CLINICAL TRIAL: NCT00248612
Title: CBT And Venlafaxine Treatments For Anxiety In Alcoholism
Brief Title: Psychosocial and Medication Treatment for Anxiety in Alcoholism
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-22529; R01AA013727-01A1 (NIH)
Record Dates: First submitted 2005-11-02; First posted 2005-11-04 (Estimated); Results first posted 2017-08-17 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Alcohol-Related Disorders; Anxiety Disorders
Keywords: Venlafaxine; Alcoholism; Anxiety Disorders; Alcohol-Use Disorders; Alcohol Abuse; Alcohol Dependence; Cognitive Behavioral Treatment
MeSH Terms: conditions — Alcohol-Related Disorders; Anxiety Disorders; Alcoholism | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Venlafaxine & CBT (Experimental): CBT is Cognitive Behavioral Treatment which will be tailored to participants. Participants will be assigned to a 12-week treatment condition; all treatment conditions will begin with a 1-week placebo run-in, after which participants will begin a trial of venlafaxine. The treatments will conclude with a 2-week medication taper.
  Interventions: Drug: Venlafaxine; Behavioral: CBT
- Placebo & CBT (Active Comparator): CBT is Cognitive Behavioral Treatment which will be tailored to participants.For patients with comorbid alcohol-use and anxiety disorders, CBT and pharmacotherapy will be contrasted with relaxation training and placebo medication; all treatment conditions will begin with a 1-week placebo run-in, after which participants will begin a trial of venlafaxine or placebo.
  Interventions: Behavioral: CBT; Other: Placebo medication
- Venlafaxine & PMR (Active Comparator): Progressive Muscle Relaxation Therapy (PMR) is a technique of alternately tensing and relaxing muscles groups in sequence throughout the body. . Participants will be assigned to a 12-week treatment condition; all treatment conditions will begin with a 1-week placebo run-in, after which participants will begin a trial. The treatments will conclude with a 2-week medication/placebo taper.
  Interventions: Drug: Venlafaxine; Other: Progressive muscle relaxation therapy (PMR)
- Placebo & PMR (Placebo Comparator): Progressive Muscle Relaxation Therapy (PMR) is a technique of alternately tensing and relaxing muscles groups in sequence throughout the body. . For patients with co-morbid alcohol-use and anxiety disorders, CBT and pharmacotherapy will be contrasted with relaxation training and placebo medication; all treatment conditions will begin with a 1-week placebo run-in, after which participants will begin a trial of venlafaxine or placebo.
  Interventions: Other: Progressive muscle relaxation therapy (PMR); Other: Placebo medication

INTERVENTIONS:
Drug: Venlafaxine — Participants will be assigned to a 12-week treatment condition; all treatment conditions will begin with a 1-week placebo run-in, after which participants will begin a trial of venlafaxine. The treatments will conclude with a 2-week medication taper.
  Other Names: Effexor XR
  Arms: Venlafaxine & CBT; Venlafaxine & PMR
Behavioral: CBT — CBT is Cognitive Behavioral Therapy. Participants will be assigned to a 12-week treatment condition; all treatment conditions will begin with a 1-week placebo run-in, after which participants will begin a trial. The treatments will conclude with a 2-week medication/placebo taper.
  Arms: Placebo & CBT; Venlafaxine & CBT
Other: Progressive muscle relaxation therapy (PMR) — For patients with comorbid alcohol-use and anxiety disorders, CBT and pharmacotherapy will be contrasted with relaxation training and placebo medication; all treatment conditions will begin with a 1-week placebo run-in, after which participants will begin a trial of venlafaxine or placebo.
  Arms: Placebo & PMR; Venlafaxine & PMR
Other: Placebo medication — For patients with comorbid alcohol-use and anxiety disorders, CBT and pharmacotherapy will be contrasted with relaxation training and placebo medication; all treatment conditions will begin with a 1-week placebo run-in, after which participants will begin a trial of venlafaxine or placebo.
  Arms: Placebo & CBT; Placebo & PMR

SUMMARY:
The proposed project is written as a "typical clinical practice" test and is a fully-controlled trial of a combined anxiety-focused CBT and pharmacotherapy (venlafaxine; CBT-VEN) delivered for patients with comorbid alcohol-use and anxiety disorders. The CBT and pharmacotherapy will be contrasted with relaxation training and placebo medication. One hundred and eighty participants will be recruited and, subsequent to a platform of outpatient treatment for alcoholism, will be randomly assigned to a 12-week treatment condition. All treatment conditions will begin with a 1-week placebo run-in, after which participants will begin a trial of venlafaxine or placebo. The treatments will conclude with a 2-week medication/placebo taper. Follow-up assessments will be conducted at post-treatment and at 3, 6, 9, and 12-months. The long-term objectives of this research are to develop a real-world combination of psychosocial and pharmacological treatments for patients with comorbid alcohol-use and anxiety disorders that compromise prognosis, and to evaluate the effectiveness of combined psychosocial and pharmacological treatments that target anxiety among patients with this comorbidity.

DETAILED DESCRIPTION:
Difficulties in anxiety management are frequent causes of relapse to alcohol use. Empirical data support the role of anxiety in alcohol relapse, and both psychosocial and pharmacological treatments for alcohol problems increasingly address the role of negative affect in alcohol-use disorders. Due to the lack of large, well-controlled treatment outcome trials, the optimal treatment (or combination of treatments) remains unknown. Real world practice in the treatment of alcohol-use disorders frequently begins with brief detoxification and stabilization, and is often followed by some combination of CBT and pharmacotherapy for patients complaining of mood difficulties while attempting early abstinence from alcohol.

The purpose of the present study is to evaluate the relative benefits of psychosocial and psychopharmacological therapy for the treatment of co-morbid anxiety and alcohol dependence among patients attempting early abstinence from alcohol. We will address the following four questions:

1. During the course of intervention, is treatment of anxiety disorders with combined treatments of established utility (among non-alcohol-use-disordered patients) superior in managing both return to drinking and anxiety symptoms than either monotherapy, or a fully inactive control treatment?
2. During the follow-up period, will patients who received the combined active treatments fare better in maintaining abstinence relative to the single active treatments, and those in the control condition?
3. What psychosocial variables (such as increases or lapses to elevated anxiety) mediate return to pre-treatment levels of alcohol use?
4. Will baseline indices of alcohol dependence and anxiety disorder severity moderate the relationship between treatment and outcome during both the acute and follow-up phases of the study?

ELIGIBILITY:
Inclusion Criteria:

* Participants must be English-speaking males or females
* Participants must be between 18 and 65 years old
* Meet criteria for DSM-IV diagnosis of alcohol abuse or dependence
* Meet criteria for Panic disorder, Social Phobia or Generalized Anxiety Disorder
* Physically able to attend sessions at the Counseling Center
* Able to read and write
* Able to complete the structured interview and self-report assessment packet
* Able to attend all treatment sessions and follow-up assessments
* Able to sign a witnessed informed consent form
* Participants express a desire to completely stop drinking alcohol or reduce alcohol consumption with the possible long-term goal of abstinence

Exclusion Criteria:

* Meet DSM-IV diagnostic criteria for bipolar disorder, schizophrenia, bulimia/anorexia, or dementia
* Currently taking anti-craving agents (e.g. Naltrexone, methadone)
* Currently taking medication that has clinically significant interactions with venlafaxine
* Previous use of venlafaxine
* Currently taking other antidepressant medications
* Currently taking medication known to decrease anxiety or alcohol consumption (e.g. antabuse)
* Currently prescribed medications with known abuse potential (e.g., subjects on opioid agonist therapy)
* Currently prescribed medications as a sleep aid (e.g. Ambien)
* Currently taking herbal supplements that have been shown to interact with venlafaxine or affect anxiety symptoms
* Currently pregnant, breastfeeding, plans of becoming pregnant during the course of the study, or not using medically acceptable form of birth control (oral contraceptives, barrier [diaphragm or condom] with spermicide, intrauterine progesterone contraceptive system, levonorgestrel implant, medroxyprogesterone acetate contraceptive injection).
* Planning to relocate out-of-state within four months of protocol initiation
* History of psychotic symptoms within the past 30 days
* Experiencing severe symptoms of depression or have engaged in suicidal behaviors within the past 30 days
* Medical contraindications to the use of venlafaxine [severe renal disease, cirrhosis, uncontrolled blood pressure, recent cardiovascular problems (e.g., heart attack), and seizure disorders; currently taking a monoamine oxidase inhibitor, MAOI]
* Self-reported anxiety less than 15 on the Hamilton Rating Scale for Anxiety
* Participant is a member of the same household of another subject already participating in the study
* Participant is legally mandated (e.g., to avoid incarceration, monetary or other penalties, etc.) to participate in an alcohol treatment program
* Participant has a current or recent (past 30 days) DSM-IV diagnosis of other substance abuse or dependence, with the exception of nicotine, marijuana, and caffeine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2003-09 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Domenic Ciraulo, MD, Principal Investigator — Boston Medical Center
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - Center for Anxiety and Related Disorders, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Following telephone screening (n=950), 162 eligible subjects completed an in-clinic baseline assessment #1 to determine eligibility for inclusion in the study.
Pre-assignment Details: Once subjects achieved the four day period of abstinence they completed a second baseline assessment in which eligibility was re-assessed. 81 Eligible subjects were then randomized into the four study arms.
Groups:
- Venlafaxine & CBT: Venlafaxine (Effexor XR): Participants will be assigned to a 12-week treatment condition; all treatment conditions will begin with a 1-week placebo run-in, after which participants will begin a trial of venlafaxine. The treatments will conclude with a 2-week medication taper. They will also receive tailored cognitive behavioral training (CBT)
- Placebo & CBT: Placebo and CBT (Cognitive Behavioral Therapy): Participants will be assigned to a 12-week treatment condition; all treatment conditions will begin with a 1-week placebo run-in, after which participants will begin a trial. The treatments will conclude with a 2-week medication/placebo taper.
- Venlafaxine & PMR: Venlafaxine and PMR (progressive muscle relaxation therapy).
- Placebo & PMR: Placebo medication and PMR (progressive muscle relaxation therapy)
Period: Overall Study
Arm/Group | Venlafaxine & CBT | Placebo & CBT | Venlafaxine & PMR | Placebo & PMR
Started | 24 | 21 | 14 | 22
Completed | 24 | 21 | 14 | 22
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Venlafaxine & CBT: Venlafaxine (Effexor XR) and CBT (Cognitive Behavioral therapy): Participants will be assigned to a 12-week treatment condition; all treatment conditions will begin with a 1-week placebo run-in, after which participants will begin a trial of venlafaxine. The treatments will conclude with a 2-week medication taper.
- Total: Total of all reporting groups
Arm/Group | Venlafaxine & CBT | Placebo & CBT | Venlafaxine & PMR | Placebo & PMR | Total
Number analyzed (Participants) | 24 | 21 | 14 | 22 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 21 | 14 | 22 | 81
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 3 | 5 | 18
  Male | 18 | 17 | 11 | 17 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21 | 18 | 12 | 19 | 70
  African American | 2 | 1 | 0 | 2 | 5
  Other | 1 | 2 | 2 | 1 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 21 | 14 | 22 | 81
Drinking status [Mean (Standard Deviation); unit: percent of days] — Drinking status was measured for the 90 day long pre-screening period by calculating the mean percent and standard deviation of the days drinking and of the days heavy drinking
  percent of days
    percent days drinking | 72.0 (24.5) | 76.0 (25.6) | 88.0 (12.7) | 76.5 (25.8) | 77 (23.8)
    percent days heavy drinking | 63.1 (28.0) | 59.1 (33.7) | 76.9 (19.1) | 67.2 (28.6) | 65.6 (28.2)
ADS Scores [Mean (Standard Deviation); unit: units on a scale] — The ADS provides a quantitative measure of the severity of alcohol dependence consistent with the concept of the alcohol dependence syndrome. The 25 items cover alcohol withdrawal symptoms, impaired control over drinking, awareness of a compulsion to drink, increased tolerance to alcohol, and salience of drink-seeking behavior. Scores range from 0-47.0= no alcohol dependence, 1-13=low, 14-21 =intermediate, 22-30= substantial and 31-47= severe level of alcohol dependence.
  units on a scale | 15.0 (7.6) | 15.8 (7.7) | 16.6 (6.6) | 16.1 (5.9) | 15.8 (7.6)
Drinks per day [Mean (Standard Deviation); unit: number of drinks] — The average number of drinks per day was obtained by taking the mean of the number of drinks each day for the 90 day long pre-screening period.
  number of drinks | 8.4 (6.5) | 7.0 (4.6) | 9.6 (4.3) | 9.7 (7.5) | 8.6 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression Scale-I (CGI-I)
Description: Global improvement of alcohol dependence: Rate the total improvement in the participant's alcohol dependence symptoms whether or not, in your judgment, it is due entirely to treatment. Compared to his/her admission to the project, how much has s/he changed?
  (1-Not assessed, first rating, 2-Very much improved, 3-Much improved, 4-Minimally improved, 5-Unchanged, 6-Minimally worse, 7-Much worse, 8-Very much worse)
Time Frame: Session 1 (Baseline) , Session 8 (8 weeks of treatment), Session 11 (11 weeks of treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Venlafaxine & CBT: Venlafaxine (Effexor XR): Participants will be assigned to a 12-week treatment condition; all treatment conditions will begin with a 1-week placebo run-in, after which participants will begin a trial of venlafaxine. The treatments will conclude with a 2-week medication taper.
- Venlafaxine & PMR; Placebo & PMR: Placebo medication and PMR (progressive muscle relaxation therapy).
Arm/Group | Venlafaxine & CBT | Placebo & CBT | Venlafaxine & PMR | Placebo & PMR
Number analyzed (Participants) | 24 | 21 | 14 | 22
units on a scale
  Session 1 CGI-I | 3.65 (1.34) | 3.81 (1.21) | 3.86 (1.10) | 4.05 (0.65)
  Session 8 CGI-I | 3.61 (1.38) | 3.13 (0.89) | 3.50 (1.09) | 3.53 (1.19)
  Session 11 CGI-I | 3.13 (1.30) | 2.61 (0.78) | 3.00 (1.15) | 2.92 (0.95)

2. Primary Outcome: Clinical Global Impression Scale-S (CGI-S)
Description: Global severity of alcohol dependence: Considering your total clinical experience with the alcohol dependent population how severe are his/her alcohol dependence symptoms at this time?
  (1-Normal, no symptoms, 2-Borderline symptoms, 3-Mild symptoms, 4-Moderate symptoms, 5-Marked symptoms, 6-Severe symptoms, 7-Among the most extreme symptoms)
Time Frame: 1 (Baseline) , Session 8 (8 weeks of treatment), Session 11 (11 weeks of treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venlafaxine & CBT | Placebo & CBT | Venlafaxine & PMR | Placebo & PMR
Number analyzed (Participants) | 24 | 21 | 14 | 22
units on a scale
  Session 1 CGI-S | 4.00 (1.24) | 3.76 (0.89) | 3.93 (0.92) | 4.18 (1.18)
  Session 8 CGI-S | 3.28 (1.49) | 2.88 (1.26) | 3.25 (1.42) | 3.40 (1.18)
  Session 11 CGI-S | 3.00 (1.88) | 2.53 (1.18) | 2.60 (1.51) | 2.85 (1.34)

3. Primary Outcome: Craving Desire Scale (CDS)
Description: The Craving Desire Scale (CDS) is a 3-item scale ("1. I do want to drink now", "2. I crave a drink right now", 3. "I have a desire for a drink right now") used to identify the degree of current alcohol craving, with responses provided on a Likert scale of 1-7: with 1 meaning strongly disagree, and 7 meaning strongly agree to each of the 3 items. Total scores can range from 3 to 21 with higher scores indicating greater craving for alcohol.
Time Frame: 1 (Baseline) , Session 8 (8 weeks of treatment), Session 11 (11 weeks of treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venlafaxine & CBT | Placebo & CBT | Venlafaxine & PMR | Placebo & PMR
Number analyzed (Participants) | 24 | 21 | 14 | 22
units on a scale
  Session 1 CDS | 8.63 (6.03) | 8.14 (5.02) | 8.21 (5.94) | 7.55 (5.06)
  Session 8 CDS | 6.44 (5.28) | 7.41 (5.06) | 4.45 (1.75) | 5.56 (3.41)
  Session 11 CDS | 4.38 (1.94) | 6.11 (4.76) | 5.10 (2.08) | 4.25 (2.70)

4. Primary Outcome: Number of Participants Abstinent
Description: Abstaining from the consumption of intoxicating beverages.
Time Frame: Session 8 (8 weeks of treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Venlafaxine & CBT | Placebo & CBT | Venlafaxine & PMR | Placebo & PMR
Number analyzed (Participants) | 24 | 21 | 14 | 22
Participants | 2 | 4 | 3 | 1

5. Secondary Outcome: Treatment Completion
Description: The number and percent of participants that completed the treatment in each arm of the study.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Venlafaxine & CBT | Placebo & CBT | Venlafaxine & PMR | Placebo & PMR
Number analyzed (Participants) | 24 | 21 | 14 | 22
Participants | 18 | 17 | 11 | 15

6. Secondary Outcome: Medication Compliance Rates
Description: The medication compliance rate is the percentage of participants in each study arm who took their medication based on pill counts.
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Venlafaxine & CBT | Placebo & CBT | Venlafaxine & PMR | Placebo & PMR
Number analyzed (Participants) | 24 | 21 | 14 | 22
percentage of participants | 96.89 | 97.06 | 88.70 | 95.39

7. Secondary Outcome: DASS Stress Subscale Score
Description: DASS (Depression Anxiety Stress Scales) assesses depression, anxiety and stress responses. Each of the three DASS scales contains 14 items, divided into subscales of 2-5 items with similar content. The stress subscale was used which assesses difficulty relaxing, nervous arousal, and being easily upset/agitated, irritable/over-reactive and impatient. Subjects are asked to use 4-point severity/frequency scales to rate the extent to which they have experienced each state over the past week. Stress scores can range form 0-56 with 0-14=normal, 15-18=mild, 19-25=moderate, 26-33=severe. and 34+=extremely severe stress.
Time Frame: Session 1 (baseline), Session 11 (11 weeks of treatment)
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venlafaxine & CBT | Placebo & CBT | Venlafaxine & PMR | Placebo & PMR
Number analyzed (Participants) | 24 | 21 | 14 | 22
units on a scale
  Session 1 DASS stress subscale | 16.7 (7.6) | 19.2 (9.1) | 21.5 (11.3) | 16.6 (8.2)
  Session 11 DASS stress subscale | 8.1 (4.6) | 9.6 (7.9) | 4.1 (7.9) | 11.2 (11.1)

8. Secondary Outcome: HAM-A Scale
Description: The Hamilton Anxiety Rating Scale (HAM-A) is a psychological questionnaire used by clinicians to rate the severity of a patient's anxiety. The HAM-A probes 14 parameters each item is scored on a 5-point scale, ranging from 0=not present to 4=severe. total scores can range from 0 to 56.where <17 indicates mild anxiety, 18-24 moderate anxiety and 25-30 severe anxiety. Higher scores reflect more anxiety.
Time Frame: Session 1 (baseline), Session 8 (8 weeks of treatment)
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venlafaxine & CBT | Placebo & CBT | Venlafaxine & PMR | Placebo & PMR
Number analyzed (Participants) | 24 | 21 | 14 | 22
units on a scale
  Session 1 HAM-A | 13.5 (5.9) | 14.2 (7.3) | 16.5 (6.8) | 12.9 (4.1)
  Session 8 HAM-A | 9.8 (6.9) | 9.1 (5.5) | 7.9 (5.5) | 9.1 (4.2)

9. Secondary Outcome: HAM-D Scale
Description: HAM-D (Hamilton Rating Scale for Depression) is a multiple item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery. The scoring is based on 17 items. Eight of the items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine items are scored on a 3 point scale from 0-2 where 0=none or absent and 2= severe. The total scores for the HAM-D can range from 0 to 50. The total scores are interpreted as: 0-7=normal, 8-13=mild, 14-18= moderate, 19-22= severe, and 23+=very severe depression. The higher the score the more severe the participant's depression.
Time Frame: Session 1 (baseline), Session 8 (8 weeks of treatment)
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Venlafaxine & CBT | Placebo & CBT | Venlafaxine & PMR | Placebo & PMR
Number analyzed (Participants) | 24 | 21 | 14 | 22
units on a scale
  Session 1 HAM-D | 12.0 (5.7) | 11.7 (6.0) | 13.0 (7.2) | 13.6 (5.0)
  Session 8 HAM-D | 8.8 (6.6) | 8.5 (4.6) | 5.9 (5.6) | 10 (6.2)

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Venlafaxine & PMR: Venlafaxine medication and PMR (progressive muscle relaxation therapy).
Arm/Group | Venlafaxine & CBT | Placebo & CBT | Venlafaxine & PMR | Placebo & PMR
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/21 | 0/14 | 0/22
Serious Adverse Events (participants affected / at risk) | 3/24 | 1/21 | 2/14 | 1/22
Other Adverse Events (participants affected / at risk) | 0/24 | 0/21 | 0/14 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venlafaxine & CBT (N=24) | Placebo & CBT (N=21) | Venlafaxine & PMR (N=14) | Placebo & PMR (N=22)
suicidal ideation (Psychiatric disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
insomnia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
agitation/restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
depression (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
elevated blood pressure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
profuse sweating (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
vertigo (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Small size of treatment groups leading to diminished meaningful difference between comparison groups at follow-up; Failure of randomization leading to unequal number of subjects in each treatment group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes